CLINICAL TRIAL: NCT03855722
Title: Remote Ischaemic Preconditioning in Transplantation (RIPTRANS) - A Prospective Randomized Controlled Trial
Brief Title: Remote Ischaemic Preconditioning in Transplantation (RIPTRANS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Finska Läkaresällskapet (funding) (Unknown); Academy of Finland (Other); Helsinki University Hospital Research Funds (funding) (Unknown)
Responsible Party: Principal Investigator, Ville Sallinen, MD, PhD, Adj. Prof., Consultant, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RIPTRANS
Record Dates: First submitted 2019-02-11; First posted 2019-02-27 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Transplant Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC (Experimental): RIPC will consist of setting a tourniquet to donor thigh and inflating it to 300mmHg four times 5 minutes with 5 minutes deflating in between each. RIPC-intervention will be performed twice: First after brain death and second time before procurement procedure.
  Interventions: Procedure: RIPC
- Sham-RIPC (Sham Comparator): Sham-RIPC will consist of setting a tourniquet to donor thigh without inflating it and keeping it in place for 35 min. Sham-RIPC-intervention will be performed twice: First after brain death and second time before procurement procedure.
  Interventions: Procedure: Sham-RIPC

INTERVENTIONS:
Procedure: RIPC — Remote Ischaemic Preconditioning
  Arms: RIPC
Procedure: Sham-RIPC — Sham procedure
  Arms: Sham-RIPC

SUMMARY:
Remote ischemic preconditioning (RIPC) is a concept where remotely induced ischemia produces protection against ischemia-reperfusion injury in a remote organ. RIPC has been studied extensively in animal models and heart surgery, but it's benefit in transplantation has been studied less. The primary aim of this study is to find out whether RIPC performed in a donor in donation after brain-death (DBD) could improve delayed graft function rate of kidney transplants.

ELIGIBILITY:
Donor Inclusion Criteria:

* Brain-dead organ donor with a plan of harvesting at least one kidney

Donor Exclusion Criteria:

* Haemodynamically unstable donor
* Age below 18 years
* Planned organ recipients are recruited to another prospective trial, which prevents participation in this trial.

All organ recipients receiving organs (kidney, liver, pancreas-kidney, heart, lungs) from a randomized donor will be recruited providing that the recipient surgery is performed at Helsinki University Hospital, recipient is over 18 years old, and recipient gives written informed consent to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2042-02 (Estimated)

PRIMARY OUTCOMES:
DGF | 7 days
  Delayed graft function of kidney allografts defined as postoperative dialysis within 1 week from transplantation

SECONDARY OUTCOMES:
Kidney allografts: eGFR | at 3 months, 1 year, 2 year, 5 year, 10 year, and 20 year
  Kidney allografts: estimated glomerular filtration rate
Combined Pancreas-Kidney allografts: eGFR | at 3 months, 1 year, 2 year, 5 year, 10 year, and 20 year
  Combined Pancreas-Kidney allografts: estimated glomerular filtration rate
Kidney allografts: BPAR | within 1 year
  Kidney allografts: Biopsy proven acute rejection
Combined Pancreas-Kidney allografts: Kidney BPAR | within 1 year
  Combined Pancreas-Kidney allografts: Biopsy proven acute rejection in Kidney allograft
Kidney allografts: graft survival | at 3 months, 1 year, 2 year, 5 year, 10 year, and 20 year
  Kidney allografts: time from transplantation to death, retransplantation or permanent dialysis
Combined Pancreas-Kidney allografts: kidney graft survival | at 3 months, 1 year, 2 year, 5 year, 10 year, and 20 year
  Combined Pancreas-Kidney allografts: time from transplantation to death, retransplantation of the kidney or permanent dialysis
Kidney allografts: death-censored graft survival | at 3 months, 1 year, 2 year, 5 year, 10 year, and 20 year
  Kidney allografts: time from transplantation to retransplantation or permanent dialysis, death-censored
Combined Pancreas-Kidney allografts: death-censored kidney graft survival | at 3 months, 1 year, 2 year, 5 year, 10 year, and 20 year
  Combined Pancreas-Kidney allografts: time from transplantation to retransplantation of the kidney or permanent dialysis, death-censored
Liver allografts: MEAF-score at 3rd POD | 3rd post-operative day
  Liver allografts: Model for Early Allograft Function Scoring (MEAF) (MEAF = (score ALTmax:3POD+ score INRmax:3POD+ score bilirubin3POD), score range 0 - 10, higher score indicates worse outcome)
Liver allografts: Postoperative biliary complications | within 1 year
  Liver allografts: Amount and type of postoperative biliary complications: stricture at anastomosis, bile leak, ischaemic type biliary lesions (ITBL)
Liver allografts: Posttransplantation kidney injury | within 1 week, at 3 months, 1 year
  Liver allografts: Posttransplantation kidney injury (acute kidney injury) according to ADQI (2010) criteria
Liver allografts: BPAR | within 1 year
  Liver allografts: Biopsy proven acute rejection
Liver allografts: graft survival | at 1 year, 2 year, 5 year, 10 year, and 20 year
  Liver allografts: graft survival: time from transplantation to death, retransplantation or explantation
Pancreas allografts: HbA1c | at 3 months, 1 year, 2 year, 5 year, 10 year, and 20 year
  Pancreas allografts: blood HbA1c measurement
Pancreas allografts: Acute rejection | within 1 year
  Pancreas allografts: Either biopsy proven (allograft pancreas or duodenal biopsy) acute rejection or clinically treated suspected acute rejection
Pancreas allografts: Pancreatic allograft survival | at 1 year, 2 year, 5 year, 10 year, and 20 year
  Pancreas allografts: Time from transplantation to death, retransplantation, explantation or daily insulin dependance
Pancreas allografts: Death-censored Pancreatic allograft survival | at 1 year, 2 year, 5 year, 10 year, and 20 year
  Pancreas allografts: Time from transplantation to retransplantation, explantation or daily insulin dependance, death-censored
Heart allograft: TnI at 6 hours | at 6 hours
  Heart allograft: blood TnI measurement at 6 hours after transplantation
Heart allograft: proBNP at 1 week | at 1 week
  Heart allograft: blood proBNP measurement at 1 week after transplantation (12/09/2019 BNP changed to proBNP because of changes in Helsinki University Hospital HUSlab laboratory protocols)
Heart allograft: Primary graft dysfunction | within 24 hours after transplantation
  Heart allograft: Primary graft dysfunction according to ISHLT (2014)
Heart allograft: acute rejection | within 1 year
  Heart allograft: Biopsy proven or clinically treated acute rejection
Heart allograft: Vasculopathy-free survival | at 1 year, 2 year, 5 year, 10 year, and 20 year
  Heart allograft: Vasculopathy-free survival according to Mehra (2010)
Heart allograft: graft survival | at 1 year, 2 year, 5 year, 10 year, and 20 year
  Heart allograft: time from transplantation to death, retransplantation or explantation
Lung allograft: Primary graft dysfunction | within 72 hours
  Lung allograft: Primary graft dysfunction according to ISHLT
Lung allograft: Acute rejection | within 1 year
  Lung allograft: Biopsy proven or clinically treated acute rejection
Lung allograft: CLAD-free survival | at 1 year, 2 year, 5 year, 10 year, and 20 year
  Lung allograft: Chronic Lung Allograft Dysfunction (CLAD) free survival according to Verleden (2014)
Lung allograft: graft survival | at 1, 2, 5, 10 and 20 year
  Lung allograft: time from transplantation to death, retransplantation or explantation (12/16/2019 secondary outcome measures for lung recipients redifined. Lung recipients recruitment started later than for other organs because of a conflicting trial which now has completed recruiting. Only four lung patients have thus far been included in the study and no results for lung recipients have been analyzed.)

OTHER OUTCOMES:
Exploratory outcomes Kidney allograft miR-21 | peroperative blood samples before and after graft perfusion and urinary sample 6 hours after transplantion
  Measurement of reperfusion injury in blood and urine samples micro-RNA miR-21
Exploratory outcomes Kidney allograft miR-24 | peroperative blood samples before and after graft perfusion and urinary sample 6 hours after transplantion
  Measurement of reperfusion injury in blood and urine samples micro-RNA miR-24
Exploratory outcomes Kidney allograft NGAL | peroperative blood samples before and after graft perfusion and urinary sample 6 hours after transplantion
  Measurement of reperfusion injury in blood and urine samples neutrophil gelatinase associated lipocain NGAL
Exploratory outcomes Kidney allograft KIM-1 | peroperative blood samples before and after graft perfusion and urinary sample 6 hours after transplantion
  Measurement of reperfusion injury in blood and urine samples kidney injury molecule -1 KIM-1
Exploratory outcomes Kidney allograft FABP-1 | peroperative blood samples before and after graft perfusion and urinary sample 6 hours after transplantion
  Measurement of reperfusion injury in blood and urine samples fatty acid binding protein -1 FABP-1
Exploratory outcomes Kidney allograft SLPI | peroperative blood samples before and after graft perfusion and urinary sample 6 hours after transplantion
  Measurement of reperfusion injury in blood and urine samples secretory leucocyte proteinase inhibitor SLPI
Exploratory outcomes Liver allograft: Early allograft dysfunction | at 7 days
  Exploratory outcomes Liver allograft: Early allograft dysfunction according to Olthoff (Bil >100, INR 1.6 or more, ALT or AST > 2000 at 7th POD
Exploratory outcomes Liver allograft: Highest ALT within 7th POD | within 7 days
  Exploratory outcomes Liver allograft: The highest ALT measurement within 7th POD
Exploratory outcomes Liver allograft: Highest INR within 7th POD | within 7 days
  Exploratory outcomes Liver allograft: The highest INR measurement within 7th POD
Exploratory outcomes Liver allograft: Highest Bil within 7th POD | within 7 days
  Exploratory outcomes Liver allograft: The highest Bil measurement within 7th POD
Exploratory outcomes heart allografts: TnI | at 1 hour, 12 hours and 24 hours
  Exploratory outcomes heart allografts: TnI measurement
Exploratory outcomes heart allografts: proBNP | at 1 day, 7 days, 14 days and 21 days
  Exploratory outcomes heart allografts: (12/09/2019 BNP changed to proBNP because of changes in Helsinki University Hospital HUSlab laboratory protocols)
Exploratory outcomes heart allografts: crea | at 1 day, 7 days, 14 days and 21 days
  Exploratory outcomes heart allografts: crea
Exploratory outcomes heart allografts: urea | at 1 day, 7 days, 14 days and 21 days
  Exploratory outcomes heart allografts: urea
Exploratory outcomes heart allografts: eGFR | at 1 day, 7 days, 14 days and 21 days
  Exploratory outcomes heart allografts: eGFR
Exploratory outcomes heart allografts: LVEF | at 1 day, 7 days, 14 days and 21 days
  Exploratory outcomes heart allografts: left ventricle ejection fraction
Exploratory outcomes heart allografts: LV wall thickness | at 1 day, 7 days, 14 days and 21 days
  Exploratory outcomes heart allografts: left ventricle wall thickness measurements
Exploratory outcomes heart allografts: tricuspidal leak | at 1 day, 7 days, 14 days and 21 days
  Exploratory outcomes heart allografts: grading of the tricuspidal valve leak
Exploratory outcomes heart allografts: Ischaemia-reperfusion injury | at 7 days, 14 days and 21 days
  Exploratory outcomes heart allografts: The appearance of ischaemia-reperfusion injury in routine biopsies
Exploratory outcomes heart allografts: fibrosis | at 7 days, 14 days and 21 days
  Exploratory outcomes heart allografts: The appearance of fibrosis associated factors in routine biopsies
Exploratory outcomes heart allografts: long time follow-up of proBNP | at 1 month, 3 months, 6 months, 12 months
  Exploratory outcomes heart allografts: long time follow-up of proBNP (12/09/2019 BNP changed to proBNP because of changes in Helsinki University Hospital HUSlab laboratory protocols)
Exploratory outcomes heart allografts: long time follow-up of LVEF | at 1 month, 3 months, 6 months, 12 months
  Exploratory outcomes heart allografts: long time follow-up of left ventricle ejection fraction in cardiac ECHO
Exploratory outcomes heart allografts: CAD at 1 year | at 1 year
  Exploratory outcomes heart allografts: Coronary Artery Disease in coronary angiography at 1 year
Exploratory outcomes heart allografts: MACE | at 1 month, 3 months, 6 months, 12 months
  Exploratory outcomes heart allografts: Major Adverse Cardiac Events (including death because of cardiac cause, graft loss, primary allograft dysfunction, rejection classified as 2R or more)
Exploratory outcomes lung allografts: Severity of ischaemia/reperfusion injury standardized P/F-ratio | at 0 hours, 1 hour, 6 hours, 12 hours and 24 hours
  Severity of ischemia/reperfusion injury after transplantation: standardized P/F-ratio during mechanical ventilation
Exploratory outcomes lung allografts: Severity of ischaemia/reperfusion injury: non-standardized P/F-ratio | at 0 hours, 1 hour, 6 hours, 12 hours and 24 hours
  Severity of ischemia/reperfusion injury after transplantation: non-standardized P/F-ratio during mechanical ventilation
Exploratory outcomes lung allografts: Severity of ischaemia/reperfusion injury: lactate | at 0 hours, 1 hour, 6 hours, 12 hours and 24 hours
  Severity of ischemia/reperfusion injury after transplantation , plasma lactate,
Exploratory outcomes lung allografts: Severity of ischaemia/reperfusion injury: CRP | at 0 hours, 1 hour, 6 hours, 12 hours and 24 hours
  Severity of ischemia/reperfusion injury after transplantation: serum highly sensitive C-reactive protein
Exploratory outcomes lung allografts: Severity of ischaemia/reperfusion injury: leuc | at 0 hours, 1 hour, 6 hours, 12 hours and 24 hours
  Severity of ischemia/reperfusion injury after transplantation blood leukocyte count
Exploratory outcomes lung allografts: Severity of ischaemia/reperfusion injury: neut | at 0 hours, 1 hour, 6 hours, 12 hours and 24 hours
  Severity of ischemia/reperfusion injury after transplantation neutrophil count
Exploratory outcomes lung allografts: FEV1 | at 1 month, 3 months, 6 months, 12 months
  Exploratory outcomes lung allografts: FEV1
Exploratory outcomes lung allografts: FVC | at 1 month, 3 months, 6 months, 12 months
  Exploratory outcomes lung allografts: FVC
Exploratory outcomes lung allografts: chronic rejection | at 1 month, 3 months, 6 months, 12 months
  Exploratory outcomes lung allografts: chronic rejection
Exploratory outcomes lung allografts: infections | at 1 month, 3 months, 6 months, 12 months
  Exploratory outcomes lung allografts: infections after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Aki Uutela, MD, Principal Investigator — Helsinki University Central Hospital; Ville Sallinen, MD, PhD, Study Director — Helsinki University Central Hospital; Marko Lempinen, MD, PhD, Study Chair — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
After the completion of the study the depersonalized data can be requested from the authors.

REFERENCES:
- [Derived] Uutela A, Helantera I, Lemstrom K, Passov A, Syrjala S, Aberg F, Makisalo H, Nordin A, Lempinen M, Sallinen V; RIPTRANS Study Group collaborators. Randomised sham-controlled double-blind trial evaluating remote ischaemic preconditioning in solid organ transplantation: a study protocol for the RIPTRANS trial. BMJ Open. 2020 Nov 16;10(11):e038340. doi: 10.1136/bmjopen-2020-038340. PMID 33199419